CLINICAL TRIAL: NCT01358825
Title: Antibody Persistence in Children Previously Vaccinated With Three Doses of Infanrix Hexa™ or Infanrix-IPV/Hib™
Brief Title: Study to Evaluate Antibody Persistence in Children Previously Vaccinated With Infanrix Hexa™ or Infanrix-IPV/Hib™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 115375; 2011-000943-26 (EudraCT Number)
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Tetanus; Poliomyelitis; Haemophilus Influenzae Type b; Acellular Pertussis; Diphtheria; Hepatitis B; Diphtheria-Tetanus-aPertussis-Poliomyelitis-Haemophilus Influenzae Type b Vaccines
Keywords: Infanrix-IPV/Hib; Long-term follow up; Persistence; Infanrix hexa
MeSH Terms: conditions — Tetanus; Poliomyelitis; Haemophilus Infections; Diphtheria; Hepatitis B | interventions — Blood Specimen Collection

ARMS (2):
- Infanrix hexa Group (Experimental): Subjects aged 5 years previously vaccinated at 3, 5 and 11 months of age with 3 doses of Infanrix hexa™ (DTPa-HBV-IPV/Hib) administered intramuscularly in study NCT00307034.
  Interventions: Procedure: Blood Sampling
- Infanrix-IPV/Hib Group (Experimental): Subjects aged 5 years previously vaccinated at 3, 5 and 11 months of age with 3 doses of Infanrix-IPV/Hib™ (DTPa-IPV/Hib) administered intramuscularly in study NCT00307034.
  Interventions: Procedure: Blood Sampling

INTERVENTIONS:
Procedure: Blood Sampling — A blood sample will be taken at 5 years of age, after vaccination in the primary study.

SUMMARY:
The aim of this study is to assess antibody persistence in infants who received three doses of Infanrix hexa™ (DTPa-HBV-IPV/Hib) or Infanrix-IPV/Hib™ (DTPa-IPV/Hib) at 3, 5 and 11 months of age in study NCT00307034.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had received 3 doses of Infanrix hexa™ or Infanrix-IPV/Hib™ in study NCT00307034.
* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) LAR(s) can and will comply with the requirements of the protocol.
* A male or female subject aged 5 years at the time of study entry.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Use of any investigational or non-registered product within 30 days prior to blood sampling.
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, polio, hepatitis B, and Hib vaccination or disease since the study NCT00307034, with the exception of hepatitis B vaccination in the DTPa-IPV/Hib group.
* Administration of immunoglobulins and/or any blood products within the 3 months prior to blood sampling.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2011-05-30 (Actual); Primary Completion 2011-07-15 (Actual); Study Completion 2011-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Norway (2):
  - GSK Investigational Site, Morvik
  - GSK Investigational Site, Oslo
- Sweden (2):
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Umeå

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=3640

REFERENCES:
- [Background] Silfverdal SA, Assudani D, Kuriyakose S, Van Der Meeren O. Immunological persistence in 5 y olds previously vaccinated with hexavalent DTPa-HBV-IPV/Hib at 3, 5, and 11 months of age. Hum Vaccin Immunother. 2014;10(10):2795-8. doi: 10.4161/21645515.2014.970494. PMID 25483640
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 115375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Infanrix Hexa Group: Subjects aged 5 years previously vaccinated at 3, 5 and 11 months of age with 3 doses of Infanrix hexa™ (administered intramuscularly) in study NCT00307034.
- Infanrix-IPV/Hib Group: Subjects aged 5 years previously vaccinated at 3, 5 and 11 months of age with 3 doses of Infanrix-IPV/Hib™ (administered intramuscularly) in study NCT00307034.
Period: Overall Study
Arm/Group | Infanrix Hexa Group | Infanrix-IPV/Hib Group
Started | 12 | 46
Completed | 12 | 45
Not Completed | 0 | 1
Not completed — Blood sample not drawn | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix Hexa Group | Infanrix-IPV/Hib Group | Total
Number analyzed (Participants) | 12 | 46 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.0 (0.0) | 5.0 (0.0) | 5.0 (0.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 3 | 32 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T).
Description: A seroprotected subject is a subject with anti-D/anti-T antibody concentrations greater than (≥) or equal to 0.1 international units per milliliter (IU/mL)
Time Frame: At Day 0
Population: The analysis was performed on the According-To-Protocol (ATP) Cohort, which included all subjects with blood sample available and who met all the eligibility criteria, complying with the procedure defined in the protocol and with no elimination code assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Infanrix-IPV/Hib Group
Number analyzed (Participants) | 12 | 45
Participants
  Anti-D | 7 | 28
  Anti-T: number analyzed (Participants) | 12 | 44
  Anti-T | 10 | 34

2. Primary Outcome: Concentrations of Antibodies Against Anti-D and Anti-T
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in milliinternational units per millilitre (mIU/mL).
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix Hexa Group | Infanrix-IPV/Hib Group
Number analyzed (Participants) | 12 | 45
IU/mL
  Anti-D | 0.13 [0.072 to 0.235] | 0.196 [0.114 to 0.338]
  Anti-T: number analyzed (Participants) | 12 | 44
  Anti-T | 0.29 [0.135 to 0.624] | 0.352 [0.207 to 0.599]

3. Primary Outcome: Number of Subjects With Anti-pertussis Toxoid (Anti-PT), Antifilamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations ≥5 ELISA Units Per Milliliter (EL.U/mL).
Description: Cut-off values assessed were greater than or equal to 5 ELISA units per millilitre (EL.U/mL) in the sera of subjects seronegative before vaccination.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Infanrix-IPV/Hib Group
Number analyzed (Participants) | 12 | 45
Participants
  Anti-PT | 0 | 9
  Anti-FHA | 12 | 41
  Anti-PRN | 8 | 34

4. Primary Outcome: Concentrations of Antibodies Against Anti-PT, Anti-FHA and Anti-PRN.
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per millilitre (EL.U/mL).
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix Hexa Group | Infanrix-IPV/Hib Group
Number analyzed (Participants) | 12 | 45
EL.U/mL
  Anti-PT | 2.5 [2.5 to 2.5] | 4.2 [2.9 to 6]
  Anti-FHA | 32.6 [11.5 to 92.5] | 50.7 [30.6 to 84.1]
  Anti-PRN | 6.2 [3.9 to 9.9] | 11.9 [8.4 to 16.8]

5. Primary Outcome: Number of Seroprotected Subjects Against Anti-hepatitis B Surface Antigen (Anti-HBs).
Description: Seroprotection = anti-HBs antibody concentration ≥ 10 milli-international units per milliliter (mIU/mL).
Time Frame: At Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group
Number analyzed (Participants) | 12
Participants | 5

6. Primary Outcome: Concentrations of Antibodies Against Anti-HBs.
Description: as for outcome 2
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Infanrix Hexa Group
Number analyzed (Participants) | 12
mIU/mL | 9 [3.9 to 20.9]

7. Primary Outcome: Number of Seroprotected Subjects Against Anti-polyribosyl Ribitol Phosphate (Anti-PRP).
Description: A seroprotected subject is a subject with anti-PRP antibody concentrations ≥ 0.15 micrograms per milliliter (μg/mL)
Time Frame: At Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Infanrix-IPV/Hib Group
Number analyzed (Participants) | 12 | 45
Participants | 10 | 40

8. Primary Outcome: Concentrations of Antibodies Against Anti-PRP.
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in micrograms per millilitre (μg/mL).
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Infanrix Hexa Group | Infanrix-IPV/Hib Group
Number analyzed (Participants) | 12 | 45
μg/mL | 0.404 [0.22 to 0.743] | 0.886 [0.558 to 1.407]

9. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: Assessed SAEs include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (up to Day 46)
Population: The analysis was performed on the Total Cohort, which included all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group | Infanrix-IPV/Hib Group
Number analyzed (Participants) | 12 | 46
Participants | 0 | 0

10. Primary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations ≥ 6.2 mIU/mL
Description: Cut-off values assessed were greater than or equal to 6.2 milliinternational units per millilitre ( mIU/mL) in the sera of subjects seronegative before vaccination.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa Group
Number analyzed (Participants) | 12
Participants | 6

ADVERSE EVENTS:
Time Frame: SAEs: during the entire study period (Day 0 to Day 46)
Description: As no vaccine was administered during the study, no safety data other than spontaneous SAEs were collected during the study.
Arm/Group | Infanrix Hexa Group | Infanrix-IPV/Hib Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/46
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.